CLINICAL TRIAL: NCT00704158
Title: A Phase I/II Study of CR011-vcMMAE in Patients With Locally Advanced or Metastatic Breast Cancer
Brief Title: Study of CR011-vcMMAE to Treat Locally Advanced or Metastatic Breast Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: CuraGen Corporation (Industry)
Responsible Party: Sponsor
Organization: Celldex Therapeutics (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR011-CLN-20
Record Dates: First submitted 2008-06-23; First posted 2008-06-24 (Estimated); Last update posted 2015-02-19 (Estimated); Status verified 2015-02

CONDITIONS: Breast Cancer
Keywords: CR011-vcMMAE; locally advanced breast cancer; metastatic breast cancer; breast cancer; CuraGen
MeSH Terms: conditions — Breast Neoplasms | interventions — CR011-vcMMAE

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: CR011-vcMMAE — administered as an intravenous infusion on Day 1 of a 21 day cycle.

SUMMARY:
This study will evaluate the safety and tolerability of CR011-vcMMAE in patients with locally advanced and metastatic breast cancer. CR011-vcMMAE will be administered intravenously (IV) once every 3 weeks (q3w) to cohorts of 3-6 patients to confirm the maximum tolerated dose (MTD) in breast cancer patients. Once the MTD is confirmed, up to 25 patients with locally advanced or metastatic breast cancer will be enrolled into the Phase II portion of the trial to further evaluate the safety and efficacy of CR011-vcMMAE.

ELIGIBILITY:
Main Inclusion Criteria:

* Females with confirmed breast cancer
* Age ≥ 18 years
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0 to 2
* Locally advanced or metastatic disease who have received at least two prior chemotherapeutic regimens for breast cancer, as follows:

  * At least one regimen must have been for locally advanced or metastatic disease
  * Subject must have received an anthracycline, a taxane, and capecitabine in any combination unless the subject was intolerant to or not a candidate for any of these agents
  * Hormonal therapy, biologic therapy (such as trastuzumab or bevacizumab), or immunotherapy do not count as one of the 2 regimens
  * Subjects with HER2/neu overexpressing tumors must have been treated with trastuzumab except in situations where the subject was intolerant to or not a candidate for trastuzumab
* Documented progressive disease within 6 months of the last regimen
* Adequate bone marrow, renal and liver function
* Signed informed consent

Main Exclusion Criteria:

* Chemotherapy, radiation, hormonal therapy, or bevacizumab within two weeks, or trastuzumab or investigational therapy within three weeks before treatment start
* Neuropathy > NCI-CTCAE Grade 1
* Active brain metastases.
* New York Heart Association class III or IV heart disease
* Unstable angina
* Uncontrolled arrhythmia
* A marked baseline prolongation of QT/QTc interval
* Pregnant or breast-feeding women, and women of childbearing age and potential who are not willing to use effective contraception

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2008-06; Primary Completion 2010-11 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of CR011-vcMMAE in breast cancer patients | throughout the study
To determine the MTD of CR011-vcMMAE in breast cancer patients | throughout the study

SECONDARY OUTCOMES:
Evaluation of efficacy (progression-free survival rate at 12 weeks, objective response rate, time to response, duration of response and time to progression) | throughout the study

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Florida Cancer Specialists, Fort Myers, Florida
  - Hematology Oncology Associates, Lake Worth, Florida
  - Georgia Cancer Specialists, Atlanta, Georgia
  - Cornell University, New York, New York
  - Tennessee Oncology, Nashville, Tennessee

REFERENCES:
- [Result] Bendell J, Saleh M, Rose AA, Siegel PM, Hart L, Sirpal S, Jones S, Green J, Crowley E, Simantov R, Keler T, Davis T, Vahdat L. Phase I/II study of the antibody-drug conjugate glembatumumab vedotin in patients with locally advanced or metastatic breast cancer. J Clin Oncol. 2014 Nov 10;32(32):3619-25. doi: 10.1200/JCO.2013.52.5683. Epub 2014 Sep 29. PMID 25267761
- See also: Phase I/II study of the antibody-drug conjugate glembatumumab vedotin in patients with locally advanced or metastatic breast cancer. — http://www.ncbi.nlm.nih.gov/pubmed/25267761